Official Title: Multimodal Pain Management After Robotic-Assisted Total Laparoscopic

Hysterectomy

NCT number: 04429022

Document Type: Informed Consent Document

Date of the Document: 11.02.2020



#### **University at Buffalo Institutional Review Board (UBIRB)**

Office of Research Compliance | Clinical and Translational Research Center Room 5018 875 Ellicott St. | Buffalo, NY 14203 UB Federalwide Assurance ID#: FWA00008824

#### Adult Consent to Participate in a Research Study

**Title of research study:** Multimodal Pain Management After Robotic-Assisted Total Laparoscopic Hysterectomy, Study 00004549

**Version Date:** 11.02.2020

Investigator: Sarah Andres, D.O.

**<u>Key Information</u>**: The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

#### Why am I being invited to take part in a research study?

You are being invited to take part in a research study because you are undergoing a robotic-assisted total laparoscopic hysterectomy.

#### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you. Regardless of whether you decide to participate, you will receive the highest level of care.
- You can ask all the questions you want before you decide.

# Why is this research being done?

The purpose of this research is to create a non-opioid pain medication regimen for robotic hysterectomies with the goal of minimizing the need for opioid pain medications after surgery. New, persistent opioid use is a common and under-recognized surgical complication which occurs in 6.5% of patients undergoing major surgery. In light of the opioid epidemic, a transition to non-opioid pain medication regimens is desired by both physicians and patients.

Non-opioid pain medications will be given before, during and after surgery. An opioid medication will be available post op for pain that is not alleviated by the non-opioid pain medication regimen (known as break-through pain). Patients will be sent home with prescriptions for non-opioid pain medications postoperatively, in addition to a small dosage of opioid medication if opioids were used while hospitalized. If patients do not use opioids postoperatively while hospitalized, they will be prescribed the non-opioid pain medication regimen. Our study will analyze opioid use in the hospital, pain scores, length of stay and return to clinic or ED for post-op pain.

# Permission to Take Part in a Human Research Study How long will the research last and what will I need to do?

We expect that you will be in this research study for one week.

You will be prescribed two medications to take by mouth once in the pre-operative area at the hospital. You will then have your hysterectomy surgery. The only change to this operation will be an injection of local pain medication into your cervix and at abdominal incision sites at the beginning of the procedure. You will receive a one-time dose of an intravenous NSAID medication called ketorolac at the end of your surgery. You will be prescribed a pain medication regimen consisting of three scheduled non-opioid pain medications and one opioid medication to take as needed for break-through pain not covered by the non-opioid pain medications. Per standard of care, you will be asked to rate your pain, on a scale from 1 to 10, by nursing staff during your hospital stay. We estimate that you will stay in the hospital for roughly one day. We include a one week duration of study because you will be prescribed a one week duration pain medication regimen to go home with.

You will be asked to take three non-opioid pain medications on a scheduled regimen. Per routine protocol, nursing staff will ask you what you pain score is while you are in the hospital recovering from your surgery.

Taking part in this research study may lead to added costs to you. At discharge, you will be prescribed gabapentin, Tylenol, celecoxib and oxycodone and you may have to pay a cost for these medications. We estimate these costs to average about \$25.00 in total. The amount you may be required to spend for your outpatient prescriptions for these medications may vary depending on your health insurance coverage.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

## Is there any way being in this study could be bad for me?

While rare, you could have an allergic reaction to any of the medications given in this study. Risk of having an adverse event to one of the below prescribed medications is also rare. Most patients taking the prescribed medications in the prescribed dosages experience few side effects.

An allergic reaction to the local anesthetic called ropivacaine is rare. Some side effects in this medication include ringing in your ears, slow or irregular heartbeat and weakness. Most patients have taken NSAIDs such as ibuprofen in the past without complication. NSAIDs taken at high doses (higher than prescribed in this study) have been associated with adverse side effects such as gastric ulcers, unusual bleeding or bruising, decreased kidney function, cough and chest pain. Similarly, most patients have taken acetaminophen in the past without complication. Acetaminophen taken at high doses (higher than prescribed in this study) have been associated with adverse side effects such as liver damage, rash, nausea, dizziness or trouble breathing. Gabapentin is a widely prescribed neuropathic medication that you may not have been prescribed before. Side effects associated with gabapentin include drowsiness and dizziness. Opioid medications will be available to you should you have pain not treated with the scheduled non-opioid pain medications. Opioid pain medications are associated with side effects including drowsiness, nausea, vomiting, respiratory depression, constipation and risk of dependence.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

# Will being in this study help me in any way?

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include a decrease in the amount of opioid medications you need to take after your

hysterectomy. You may also have improved pain control after surgery. Improved pain control may help you minimize the time you spend admitted to the hospital after your surgery and minimize your risk of opioid dependence.

#### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You may choose not to enroll in this study. Instead of being in this research study, your choices include having a traditional pain medication regimen after a hysterectomy. You would not have local anesthetics injected into your cervix or at abdominal incision sites. Non-opioid pain medications may or may not be scheduled. You may be prescribed a higher dose of opioid pain medications.

**Detailed Information:** The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team. The research team's contact information has been listed below:

Dr. Sarah Andres, D.O., Principal Investigator

P: (774) 451-5695

E: seandres@buffalo.edu

Dr. George Danakas, M.D.

P: (716) 883-4350

E: gdanakas@gppconline.com

Dr. Armen Kirakosyan, M.D.

P: (716) 656-4077

E: akirakosyan@kaleidahealth.org

You may also contact the research participant advocate at 716-888-4845 or researchadvocate@buffalo.edu.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). An IRB is a committee that provides ethical and regulatory oversight of research that involves human subjects. You may talk to them at (716) 888-4888 or email <a href="mailto:ub-irb@buffalo.edu">ub-irb@buffalo.edu</a> if:

- You have questions about your rights as a participant in this research
  - Your questions, concerns, or complaints are not being answered by the research team.
  - You cannot reach the research team.
  - You want to talk to someone besides the research team.
  - You want to get information or provide input about this research.

# How many people will be studied?

We expect about 200 people will be in this research study in the Kaleida Health System in Buffalo.

# What happens if I say yes, I want to be in this research?

- You will be asked to have two blood tests (a complete blood count (CBC) and a complete metabolic panel (CMP)) completed prior to your hysterectomy. No blood samples will be retained for this research. Obtaining CBC and CMP results are routine prior to a hysterectomy and are the standard of care.
- On the day of your hysterectomy, you will be given two medications, acetaminophen and gabapentin, to take by mouth in the pre-operative area. You will not need to arrive earlier to the pre-operative area.
- After you go to sleep for your hysterectomy, a surgeon will inject a local anesthetic called ropivacaine into your cervix. Ropivacaine will also be injected at the small abdominal incisions on your abdomen.
- Your hysterectomy will be completed robotically, as planned.
- At the end of the procedure before you wake up, you will be given a dose of intravenous NSAID medication called ketorolac. Ketorolac is a medication that is routinely used after a hysterectomy and other surgeries.
- For pain management after your surgery, you will be prescribed acetaminophen, gabapentin and celecoxib by mouth on a scheduled regimen. You will be prescribed gabapentin and celecoxib to take every 12 hours for seven days. You will be prescribed acetaminophen to take every six hours for the first two days after your surgery, then as needed afterwards. You will be given these medications while in the hospital and will be prescribed them to take when you are discharged.
- You will also have an intravenous opioid medication called hydromorphone to use as needed for breakthrough pain. If you are in severe pain, you should ask your nurse for this medication.
- Per standard of care, you will be asked to rate your pain, on a scale from 1 to 10, by nursing staff during your hospital stay.
- You will have standard medications we give after a hysterectomy to treat any nausea, vomiting or gas pains that you may have.
- A complete blood count will be obtained while you are in the hospital after your surgery to measure if you have a drop in hemoglobin. This again is standard of care.
- If you need hydromorphone for pain management while you are staying in the hospital, we will additionally send a prescription for oxycodone (a similar opioid medication that can be taken by mouth) to your pharmacy. Again, we recommend you take this medication only if needed for breakthrough pain not covered by the gabapentin, celecoxib and acetaminophen medication regimen. If you do not need any opioid medications while you are in the hospital, we will only send prescriptions for acetaminophen, gabapentin and celecoxib to your pharmacy. We encourage you to call the Dr Danakas or Dr Kirakosyan if this pain medication regimen does not treat your pain adequately.
- You will have a routine post-operative appointment with your surgeon two weeks after your hysterectomy. This again is standard of care.

# What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for taking prescribed medications on a schedule after your hysterectomy.

# Permission to Take Part in a Human Research Study What happens if I say yes, but I change my mind later?

You can leave the research at any time it will not be held against you.

If you decide to leave the research, contact the investigator so that the investigator can ensure that your pain is treated adequately and we ensure documentation of any adverse events if they have occurred.

If you wish to terminate your participation in the research, previously collected data may not be removed from the study database. You will be asked whether the investigator can collect data from your routine medical care. [Note: Studies with FDA-regulation cannot have data removed from the study.] If you agree, this data will be handled the same as research data. [Note: If a subject withdraws from the interventional portion of a study and does not consent to continued follow-up of associated clinical outcome information, the investigator must not access for purposes related to the study the subject's medical record or other confidential records requiring the subject's consent. However, an investigator may review study data related to the subject collected prior to the subject's withdrawal from the study, and may consult public records, such as those establishing survival status.]

# Is there any way being in this study could be bad for me? (Detailed Risks)

While rare, you could have an allergic reaction to any of the medications given in this study. Risk of having an adverse event to one of the below prescribed medications is also rare. Most patients taking the prescribed medications in the prescribed dosages experience few side effects. NSAIDs, acetaminophen and opioid medications are considered part of the standard of care for pain management after a hysterectomy. Local anesthetics for pain are also widely used and well tolerated.

Gabapentin, while commonly used for post-operative pain control, is not officially FDA approved for this indication. Taking Gabapentin in addition to opioid medications may result in greater drowsiness or even respiratory depression. It will be very important to follow the instructions on the use of these medications at the time you are discharged from the hospital. If you have any questions about using these medications together, you should contact the PI, Dr. Sarah Andres.

An allergic reaction to the local anesthetic called ropivacaine is rare. Some side effects in this medication include ringing in your ears, slow or irregular heartbeat and weakness. Most patients have taken NSAIDs such as ibuprofen in the past without complication. NSAIDs taken at high doses (higher than prescribed in this study) have been associated with adverse side effects such as gastric ulcers, unusual bleeding or bruising, decreased kidney function, cough and chest pain. Similarly, most patients have taken acetaminophen in the past without complication. Acetaminophen taken at high doses (higher than prescribed in this study) have been associated with adverse side effects such as liver damage, rash, nausea, dizziness or trouble breathing. Gabapentin is a widely prescribed neuropathic medication that you may not have been prescribed before. Side effects associated with gabapentin include drowsiness and dizziness. Opioid medications will be available to you should you have pain not treated with the scheduled non-opioid pain medications. Opioid pain medications are associated with side effects including drowsiness, nausea, vomiting, respiratory depression, constipation and risk of dependence.

You and your insurance company will be charged for the health care services that you would ordinarily be responsible to pay. In some cases, insurance will not pay for services ordinarily covered because these services were performed in a research study. You should check with your insurance to see what services will be covered by your insurance and what you will be responsible to pay.

Breach of confidentiality is always a risk however collected information in this study is generally benign. Assigning a number to each record in the spreadsheet and coding the record will minimize it risk for breach of confidentiality.

## What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical or education records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the University at Buffalo IRB and other representatives of this organization such as the Food and Drug Administration.

If personal identifiers are removed from your identifiable private information that is collected during this research, that information could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent. This de-identified data will be stored in a datasheet that is password encrypted, on a UB domain that is also password security protected with two-factor authentication sign in. Only the research team will have access to the password protected spreadsheet.

The sponsor, monitors, auditors, the IRB, the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Federal law provides additional protections of your medical records and related health information. These are described in the HIPAA section of this document.

# Can I be removed from the research without my OK?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include inability to take or an adverse event to the study medications.

We will tell you about any new information that may affect your health, welfare, or choice to stay in the research.

#### What else do I need to know?

#### What medical costs am I responsible for paying?

The procedures and medications required by the research study that would not otherwise be part of your standard care will not be covered by the sponsor of this study. The tests or procedures that would be provided to any patient with your condition, regardless of whether he/she was participating in the research study, are considered standard care and will be billed to you or your private or public health insurance company. You will still be responsible for the cost of your usual ongoing medical care, including deductibles and co-payments. If you have any questions about what expenses are covered by the sponsor and what expenses are the responsibility of you or your health insurance provider, please contact a member of the study staff and/or your health insurance provider.

#### Who will pay for my medical care if participating in this research harms me?

It is important that you tell your study doctor if you feel that taking part in this study has injured you or caused you to become ill.

You will receive medical treatment if you are injured or become ill as a result of this study. Your doctor will explain the treatment options to you and tell you where you can get treatment.

The University at Buffalo and Kaleida Health makes no commitment to provide free medical care or payment for any unfavorable outcomes that result from your participation in this research. Medical services will be billed at the usual charge and will be your responsibility or that of your third-party payer but you are not precluded from seeking to collect compensation for injury related to malpractice, fault, or blame on the part of those involved in the research including Kaleida Health and the University at Buffalo.

By accepting medical care or accepting payment for medical expenses, you are not waiving any of your legal rights.

#### Will I get paid for my participation in this research?

You will not be paid for participating in this study.

#### What are my alternatives to participating in this research study?

KALEIDA Health, Buffalo NY

Principal Investigator

Instead of being in this research study, your choices may include: standard post-operative pain control management. Most patients will take a combination of medications including ketorolac, ibuprofen, acetaminophen and opioids. The important risks and possible benefits of these alternatives include a possible increase in opioid medication usage.

#### What will happen to my information?

Your information will be de-identified. The de-identified information will be aggregated and may be published with the goal of improving care practices for patients in the future. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

# HIPAA: Authorization for the Use and Disclosure of Identifiable Health Information for Research Purposes

This section describes information about you and about your health that will be obtained by the researchers when you participate in the research study. By signing this form, you are agreeing to permit the researchers and/or other parties (described in detail below) to have access to this information and to use or disclose it for the purposes of the research described in this document. If there are any parts of this form that you do not understand, please be sure to ask us for further clarification

# A. What individually identifiable health information will be collected about you as part of this research study? √ Information from your full medical records: age, body mass index (BMI), smoking status, prior pelvic surgeries, preinvasive or benign vs malignant disease diagnosis, history of diabetes, history of substance use disorder, pre-operative blood glucose level, pre-operative blood albumin level, operation time, blood loss during operation, post-operative hemoglobin, intraoperative complications, whether cancer staging was performed, opioid use after surgery, pain scores, length of stay in hours and return to the clinic or emergency department due to postoperative pain within a two week period. B. Who is authorized to create or provide this information for research use?

| C. Who is authorized to receive the information from the information providers identified in (B)? |
|---|
| $\underline{\hspace{0.1cm}}^{\hspace{0.1cm}}\underline{\hspace{0.1cm}}^{\hspace{0.1cm}}$ Principal Investigator or designee |
| D. With whom may your protected health information be shared? |
| Your health information may be shared with others outside of the research group for purposes directly related to the conduct of this research study or as required by law, including but not limited to: |
| Clinical staff not involved in this research study who may become involved in your care if it is potentially relevant to your treatment |
| Your information may also be shared with individuals or entities responsible for general administration, oversight and compliance of research activities. Examples of this include the institution's Privacy and Security Officers or other internal oversight staff, Safety Monitoring Boards, an Institutional Review Board, The Research Foundation of the State University of New York, University at Buffalo Foundation Services, and accrediting bodies, or with certain government oversight agencies that have authority over the research including the Department of Health and Human Services (HHS), the Food and Drug Administration (FDA), the National Institutes of Health (NIH), and the Office of Human Research Protections (OHRP). Your information may also be shared with other entities as permitted or required by law. All reasonable efforts will be used to protect the confidentiality of your individually identifiable health information that may be shared with others as described above. |
| Although safeguards are in place to prevent accidental disclosure of your information beyond the purposes described above, the information disclosed through this authorization is no longer protected by HIPAA. There is the potential for this information to be re-disclosed by the recipient(s). After such a disclosure, the information may no longer be protected by the terms of this authorization against further re-disclosure. |
| E. How long are the information providers listed in (B) authorized to provide your information for this research project? |
| $\underline{}$ b. This authorization will expire at the end of the research study. After that time, this authorization may not be used to acquire additional information about you. |
| d. Your protected health information will go into a database that will be maintained indefinitely. Any future study using this information that falls outside the scope of this current study will be required to follow guidelines designed to govern access to that information and to protect the privacy of that information. The researchers may |

#### F. What are your rights after signing this authorization?

you unless you revoke this authorization in writing.

You have the right to revoke this authorization at any time. If you withdraw your authorization, no additional efforts to collect individually identifiable health information about you will be made. You should know, however, that protected health information acquired using this

continue to rely on this authorization to acquire protected health information about

authorization prior to its withdrawal may continue to be used to the extent that the investigator(s) have already relied on your permission to conduct the research. If you chose to withdraw this authorization, you must do so in writing to the following individual:

Dr. Sarah Andres, D.O., Principal Investigator

E: seandres@buffalo.edu

A: Conventus, 5<sup>th</sup> floor, Obstetrics & Gynecology Department 1001 Main Street Buffalo, NY 14203

If you send us a request to withdraw your authorization, we will forward that request to the institutions we have shared it with in order to collect your individually identifiable health information.

#### G. What will happen if you decide not to sign this authorization?

Refusing to sign this authorization will not affect the present or future care you receive at this institution and will not cause any penalty or loss of benefits to which you are otherwise entitled. If you decide not to sign this authorization, you will not be able to participate in the research study.

Should you agree to participate in this research, this consent document will be placed in your medical record.

#### Signature Block for Capable Adult

Your signature documents your permission to take part in this research. By signing this form, you

| are not waiving any of your legal rights, including the right to seek to negligence or misconduct of those involved in the research. | compensation for injury related |
|---|---|
| Signature of subject | Date |
| Printed name of subject | |
| Signature of person obtaining consent | Date |
| Printed name of person obtaining consent | |